CLINICAL TRIAL: NCT04382768
Title: Extended Compassionate Use Program (UCA) With Inhalational Ibuprofen in Patients With Acute Respiratory Pathology, Mediated by COVID-19.
Brief Title: Inhaled Ibuprofen to Treat COVID-19
Acronym: CórdobaTrail
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Química Luar SRL (Industry)
Collaborators: National Council of Scientific and Technical Research, Argentina (Other Government); Centro de Excelencia en Productos y Procesos Córdoba (Unknown)
Responsible Party: Principal Investigator, Néstor H García, Principal Investigator, National Council of Scientific and Technical Research, Argentina
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DNL000004
Record Dates: First submitted 2020-05-06; First posted 2020-05-11 (Actual); Last update posted 2020-06-11 (Actual); Status verified 2020-06

CONDITIONS: Coronavirus Infection; Respiratory Disease; SARS (Disease)
MeSH Terms: conditions — Coronavirus Infections; Respiration Disorders; Severe Acute Respiratory Syndrome; Disease

STUDY DESIGN:
Intervention Model Description: This is an expanded compassionate use program for patients infected with SARS-CoV-2. All patients or their legally authorized representative must provide written informed consent and the patient will be examined to assess their eligibility. Eligible patients will receive inhalation ibuprofen ate three times a day, plus standard care, until the patient became negative, or their physician considers enough or the patient requested to stop.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Luarprofen (Experimental): Inhaled Hypertonic ibuprofen 50 mg tid
  Interventions: Drug: Inhaled Hypertonic ibuprofen

INTERVENTIONS:
Drug: Inhaled Hypertonic ibuprofen — Standard of care plus lipid ibuprofen 50mg tid

SUMMARY:
The study aims to evaluate the reduction in severity and progression of lung injury with inhaled ibuprofen in patients with severe acute respiratory syndrome due to SARS-CoV-2 virus.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent by the patient OR by the patient's Legal Representative.
2. Confirmed or suspected SARS-CoV-2 infection;
3. Pneumonia without criteria of severity.
4. With some of the following conditions:

   * Diabetes.
   * Cardiovascular disease.
   * Chronic kidney disease.
   * Chronic obstructive pulmonary disease.
   * Structural diseases of the lung
   * Immunocompromise.
5. Patient who presents negative results by rtPCR for SARS CoV-2, in case of being highly suspicious, the patient may receive it empirically until the results are obtained.
6. No unstable bronchial asthma

Exclusion Criteria:

1. The doctor considers that participation in the Program is not the best for patients or for any condition that prevents the Program from being followed safely.
2. Patients with a history of unstable bronchial asthma
3. The patient is allergic to ibuprofen or any of the compounds in the preparation.
4. Hypersensitivity to the drug, nasal polyps syndrome, angioedema or bronchospasm against aspirin or other NSAIDs.
5. Pregnant or lactating woman, or positive pregnancy test on a pre-dose exam.
6. Patient who is expected to be transferred to another place other than the place where the Program starts, within 7 days of starting it.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-05-01 (Actual); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Change in the scale of ordinary COVID results at 7, 14 and 28 days in patients with acute respiratory infection, induced by SARS-CoV-2, treated with inhaled Ibuprofen. | 7, 14 and 28 days
  Time to clinical improvement: defined as time from inhaled Ibuprofen first dose to an improvement of three points from the status on a seven-category ordinary scale
Change to Negativization of the swab to the following treatment points on day 7, day 14, 21 and 28 after treatment with inhaled Ibuprofen. | 7, 14 and 28 days
  Negativization of two consecutive pharyngo-nasal swab 24-72 hrs apart

SECONDARY OUTCOMES:
Chage in length of Hospital stay | 28 days
Chage in duration of ventilation | 28 days
Chage in length of Critical Care stay | 28 days
Average score of National Early Warning (NEWS2) between days 1, 7, 14 and 28. | 1, 7, 14 and 28
  NEWS2 score 20 points is the maximum and indicates that the patient needs emergent assessment by a clinical team or critical care team and usually transfer to higher level of care.
Average change in quick sepsis-related organ failure assessment score (qSOFA) score between day 1, 7, 14 and 28. | 1, 7, 14 and 28 days
  qSOFA, score for sepsis, a maximum value of 3 indicates high risk qSOFA Scores 2-3 are associated with a 3- to 14-fold increase in in-hospital mortality. Assess for evidence of organ dysfunction with blood testing including serum lactate and calculation of the full SOFA Score.
  Patients meeting these qSOFA criteria should have infection considered even if it was previously not.
Time from first dose to conversion to normal or mild pneumonia | 28 days
Antibiotic requirement | 28 days
Glucocorticoids requirement | 28 days
Incidence of adverse event | 28 days
Incidence of serious adverse event | 28 days
Number of deaths from any cause at 28 days | 28 days
Lymphocyte count | 28 days

CONTACTS AND LOCATIONS:
Overall Officials: Dante M Beltramo, PhD, Study Director — Centro de Excelencia en Productos y Procesos Córdoba
Locations (1):
- Centro de Excelencia en Productos y Procesos Córdoba, Córdoba, Argentina

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Munoz AJ, Alasino RV, Garro AG, Heredia V, Garcia NH, Cremonezzi DC, Beltramo DM. High Concentrations of Sodium Chloride Improve Microbicidal Activity of Ibuprofen against Common Cystic Fibrosis Pathogens. Pharmaceuticals (Basel). 2018 May 17;11(2):47. doi: 10.3390/ph11020047. PMID 29772761
- [Result] He L, Ding Y, Zhang Q, Che X, He Y, Shen H, Wang H, Li Z, Zhao L, Geng J, Deng Y, Yang L, Li J, Cai J, Qiu L, Wen K, Xu X, Jiang S. Expression of elevated levels of pro-inflammatory cytokines in SARS-CoV-infected ACE2+ cells in SARS patients: relation to the acute lung injury and pathogenesis of SARS. J Pathol. 2006 Nov;210(3):288-97. doi: 10.1002/path.2067. PMID 17031779
- [Result] Veljkovic V, Vergara-Alert J, Segales J, Paessler S. Use of the informational spectrum methodology for rapid biological analysis of the novel coronavirus 2019-nCoV: prediction of potential receptor, natural reservoir, tropism and therapeutic/vaccine target. F1000Res. 2020 Jan 27;9:52. doi: 10.12688/f1000research.22149.4. eCollection 2020. PMID 32419926
- [Derived] Salva O, Doreski PA, Giler CS, Quinodoz DC, Guzman LG, Munoz SE, Carrillo MN, Porta DJ, Ambasch G, Coscia E, Diaz JLT, Bueno GD, Fandi JO, Maldonado MA, Pena Chiappero LE, Fournier F, Perez HA, Quiroga MA, Sala Mercado JA, Martinez Picco C, Beltran MA, Arganaras LA, Rios NM, Kalayan GI, Beltramo DM, Garcia NH. Reversal of SARS-CoV2-Induced Hypoxia by Nebulized Sodium Ibuprofenate in a Compassionate Use Program. Infect Dis Ther. 2021 Dec;10(4):2511-2524. doi: 10.1007/s40121-021-00527-2. Epub 2021 Aug 30. PMID 34460083